CLINICAL TRIAL: NCT05424276
Title: A Phase 2 Study of IkT-148009 in Untreated Parkinson's Disease
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Trial of IkT-148009 in Untreated Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ABLi Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IkT-148009-201
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Untreated Parkinsons disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 50mg IkT-148009 (risvodetinib) (Experimental): This arm consisted of participants treated with the 50mg dose of risvodetinib.
  Interventions: Drug: IkT-148009 (risvodetinib)
- 100mg IkT-148009 (risvodetinib) (Experimental): This arm consisted of participants treated with the 100mg dose of risvodetinib.
  Interventions: Drug: IkT-148009 (risvodetinib)
- 200mg IkT-148009 (risvodetinib) (Experimental): This arm consisted of participants treated with the 200mg dose of risvodetinib.
  Interventions: Drug: IkT-148009 (risvodetinib)
- Placebo (Placebo Comparator): This arm consisted of participants treated with placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IkT-148009 (risvodetinib) — Oral administration gelatin capsule
  Arms: 100mg IkT-148009 (risvodetinib); 200mg IkT-148009 (risvodetinib); 50mg IkT-148009 (risvodetinib)
Drug: Placebo — Oral administration gelatin capsule
  Arms: Placebo

SUMMARY:
This study investigates the safety and tolerability of drug IkT-148009 in untreated Parkinson's disease volunteers (30 to 80 years old). It also looks at the pharmacokinetics of IkT-148009 in the body and evaluates the effect of IkT-148009 on motor and non-motor features of the disease. This 12 week study is designed to be 3:1 randomized across 3 doses of IkT-148009 or placebo. Each participant will self-administer one of 3 doses or placebo of IkT-148009 once daily (QD) with food for 12 weeks. For more information, visit our website: www.the201trial.com

DETAILED DESCRIPTION:
This is a 12-Week, randomized, double-blind, multi-center, placebo-controlled dose-ranging clinical trial of three IkT 148009 doses in patients with untreated PD designed to assess safety, tolerability, and pharmacokinetics of IkT-148009, an oral, once daily c-Abl tyrosine kinase inhibitor. Secondary and exploratory assessments will evaluate the effect of IkT-148009 on motor and non-motor features of the disease. 120 participants are anticipated to be enrolled at up to 34 sites across the US.

Participants will undergo screening to evaluate their eligibility to participate in the study to include evaluation of Parkinson's diagnosis, vital signs, blood chemistry, hematology and urinalysis and complete listing of concomitant medications. An Enrollment Authorization Committee (EAC) will be responsible for reviewing screening data and confirming the eligibility and suitability of participants. Those selected will be enrolled and randomized to one of three active IkT-148009 arms (50/100/200 mg) or a placebo arm (1:1:1:1). All clinical staff, study investigators, and participants will be blinded to study assignments throughout the trial.

A Data Safety Monitoring Committee (DSMB) will evaluate all available safety, tolerability, and PK and Parkinson's disease-related data for each cohort on a monthly to quarterly basis. Adverse event reporting will be evaluated in real-time.

ELIGIBILITY:
Inclusion Criteria

1. Participants who are diagnosed with PD consistent with UK Brain Bank criteria and MDS Research Criteria; must include bradykinesia with sequence effect and motor asymmetry.
2. Receiving no anti-parkinsonian therapy
3. Modified Hoehn/Yahr Stage < 3.0
4. Montreal Cognitive Assessment ≥ 24
5. Patient expected to be able to participate in trial without need for additional anti-parkinsonian therapy

Sex and Contraceptive/Barrier Requirements:

1. Male participants must agree to practice an acceptable method of highly effective birth control from the screening visit, while on study and for 30 days after receiving the last dose of study drug. Highly effective methods of birth control include sexual abstinence, vasectomy, or a condom with spermicide (men) in combination with their partner's highly effective method.
2. Female participants of childbearing potential and male participants with female partners of childbearing potential must agree to either remain abstinent or use adequate and reliable contraception throughout the study and at least 30 days after the last dose of study drug has been taken.

Informed Consent:

1. Capable of giving signed ICF as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Other Inclusions:

1. Approved as an appropriate and suitable candidate by the EAC.

Exclusion Criteria

1. Diagnosis/suspicion of secondary or atypical parkinsonism
2. Previous procedure or surgery for PD, or anticipation of these during the study
3. High likelihood of needing anti-parkinsonian treatment over the study period, in the opinion of the investigator
4. Clinically significant orthostatic hypotension
5. Clinically significant hallucinations requiring antipsychotic use in the 12 months prior to Screening
6. Clinically significant medical, surgical, psychiatric, or laboratory abnormalities in the judgement of the treating investigator or the EAC

Prior/Concomitant Therapy:

1. Past treatment with levodopa, dopaminergic agonists, monoamine oxidase-B inhibitors, supplements containing levodopa (i.e. Mucana pruriens), or A2A antagonists for more than 28 days, or treatment with any of these medications or supplements within 28 days prior to screening
2. Past treatment with irreversible monoamine oxidase-B inhibitors (e.g., selegiline) for more than 28 days; must be discontinued for at least 90 days before screening
3. Currently receiving moderate or strong Cytochrome P450 (CYP) 3A4/5 inducers or CYP3A4/5 inhibitors (except for topical administration)
4. Currently receiving any antipsychotic, metoclopramide, reserpine, or amphetamine.

Prior/Concurrent Clinical Study Experience:

1. Current participation in another investigational clinical trial and/or receipt of any investigational medication within 90 days prior to screening
2. Previous randomization into this or another IkT-148009 study

Diagnostic Assessments:

1. Active suicidal ideation within one year prior to screening visit, as determined by the Columbia Suicide Rating Scale (answer of "yes" on question 4 or 5)
2. Current diagnosis or history of substance abuse (excluding nicotine or caffeine) by Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria
3. Medical or recreational use of marijuana in the 3 months prior to the screening visit
4. Any social or behavioral reason that would preclude completion of the study, in the judgement of the investigator
5. Any skin condition that would interfere with obtaining adequate samples
6. Evidence of advanced, age-related macular degeneration (neovascular or geographic atrophy) or intermediate macular degeneration as defined by Beckman classification (Large drusen > 125 um and/or any AMD pigmentary abnormalities). Evidence of retina/choroid neovascularization from any cause. Evidence of central serous retinopathy.
7. Abnormal amylase and/or lipase at screening (may be repeated during screening period)
8. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 2.5 times the upper limit of normal (ULN)
9. Significant renal impairment as determined by the following criteria:

   * Creatinine clearance (CrCL) less than or equal to 60 mL/min for subjects < 65 years of age
   * Creatine clearance (CrCL) greater than or equal to 55 mL/min and the absence of proteinuria or hematuria for subjects ≥ 65 years of age
10. Currently lactating, pregnant or planning on becoming pregnant during the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2025-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milton Werner, PhD, Principal Investigator — ABLi Therapeutics, Inc.
Locations (27):
- United States (27):
  - Neurology, Scottsdale, Arizona
  - Neurology, Little Rock, Arkansas
  - Neurology, Reseda, California
  - Neurology, Stamford, Connecticut
  - Neurologist, Boca Raton, Florida
  - Neurology, Miami, Florida
  - Neurology, Naples, Florida
  - Neurology, Tampa, Florida
  - Neurology, Foxborough, Massachusetts
  - Neurology, South Dartmouth, Massachusetts
  - Neurology, Farmington Hills, Michigan
  - Neurology, Golden Valley, Minnesota
  - Neurology, West Long Branch, New Jersey
  - Neurology, Durham, North Carolina
  - Neurology, Raleigh, North Carolina
  - Neurology, Columbus, Ohio
  - Neurology, Tulsa, Oklahoma
  - Neurology, Portland, Oregon
  - Neurology, Port Royal, South Carolina
  - Neurology, Memphis, Tennessee
  - Neurology, Nashville, Tennessee
  - Neurology, Frisco, Texas
  - Neurology, Houston, Texas
  - Neurology, Round Rock, Texas
  - Neurology, Kirkland, Washington
  - Neurology, Madison, Wisconsin
  - Neurology, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: End of study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 32 clinical sites in the United States including both private clinics and public institutions. A total of 137 participants were enrolled in the study.
Groups:
- 50mg IkT-148009 (Risvodetinib): This arm consisted of participants treated with the 50mg dose of risvodetinib for 12 weeks.
- 100mg IkT-148009 (Risvodetinib): This arm consisted of participants treated with the 100mg dose of risvodetinib for 12 weeks.
- 200mg IkT-148009 (Risvodetinib): This arm consisted of participants treated with the 200mg dose of risvodetinib for 12 weeks.
- Placebo: This arm will consist participants treated with placebo for 12 weeks.
Period: Overall Study
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Started | 35 | 34 | 33 | 35
Completed | 31 | 31 | 28 | 30
Not Completed | 4 | 3 | 5 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Subjects Withdrawn due to regulatory hold | 3 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo | Total
Number analyzed (Participants) | 35 | 34 | 33 | 35 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.79) | 63.3 (8.08) | 63.2 (7.41) | 64.9 (7.20) | 63.7 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 11 | 16 | 55
  Male | 23 | 18 | 22 | 19 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 32 | 31 | 32 | 34 | 129
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 0 | 5 | 14
  Not Hispanic or Latino | 29 | 31 | 33 | 29 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Hoehn & Yahr [Count of Participants; unit: Participants] — Clinician's assessment of a particiapnt's disease severity at the time of screening. The scale is based on a rating of 0-5 with 0 representing no signs of disease and 5 representing a participant that is wheelchair bound or bedridden.
  Participants
    H&Y 2.5 | 0 | 1 | 0 | 2 | 3
    H&Y 2.0 | 20 | 21 | 27 | 25 | 93
    H&Y 1.5 | 2 | 1 | 3 | 0 | 6
    H&Y 1.0 | 13 | 9 | 2 | 8 | 32
    Missing | 0 | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Secondary Outcome: LS Mean of Change From Baseline in MDS-UPDRS Part II+III From a Mixed Model for Repeated Measures
Description: Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Parts II and III reflect assessments covering activites of daily living as reported by the participant (Part II) as well as a clinicians assessment of motor abilities (Part III). Part II consists of 13 items with total scores ranging from 0 to 52 while Part III consists of 18 items with total scores range from 0 to 132. Each item is scored 0 (normal) to 4 (severe). The sum of Parts 2 and 3 have a score range of 0 to 184 (31 total items). An increase in sum of Parts 2 and 3 relative to baseline represents a worsening of the participant's Parkinson's disease
Time Frame: Baseline to Week 12
Population: The mITT population will include all randomized participants who have a valid baseline MDS-UPDRS, received at least one dose of study drug, and have at least one post-baseline evaluation of the MDS-UPDRS assessment as defined in the Statistical Analysis Plan
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on the Scale
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Score on the Scale | 0.08 [-2.585 to 2.745] | 1.82 [-0.794 to 4.433] | 2.12 [-0.627 to 4.871] | 0.85 [-1.791 to 3.488]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo from baseline to 12 weeks of treatment; Test type: Superiority; p = 0.686, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.77, 95% CI 2-sided [-4.522 to 2.985], Standard Error of Mean 1.895
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo from baseline to 12 weeks of treatment; Test type: Superiority; p = 0.606, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.97, 95% CI 2-sided [-2.745 to 4.687], Standard Error of Mean 1.876
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo from baseline to 12 weeks of treatment; Test type: Superiority; p = 0.509, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 1.27, 95% CI 2-sided [-2.539 to 5.086], Standard Error of Mean 1.925

2. Secondary Outcome: LS Mean of Change From Baseline in PDQ-39 From a Mixed Model for Repeated Measures
Description: Parkinson's Disease Questionnaire (PDQ) consists of 39 questions evaluating activities of daily living. Participants rate each question on a 5 point scale (0 to 4), . The PDQ-39 score ranges from 0 to 100 with higher score representing more advanced disease.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment Score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment Score | -1.90 [-3.434 to -0.364] | -0.99 [-2.494 to 0.515] | -1.89 [-3.478 to -0.308] | -2.35 [-3.868 to -0.824]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo after 12 weeks of treatment; Test type: Superiority; p = 0.683, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.45, 95% CI 2-sided [-1.717 to 2.611], Standard Error of Mean 1.093
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo after 12 weeks of treatment; Test type: Superiority; p = 0.212, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 1.36, 95% CI 2-sided [-0.783 to 3.495], Standard Error of Mean 1.080
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo after 12 weeks of treatment; Test type: Superiority; p = 0.685, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.45, 95% CI 2-sided [-1.749 to 2.654], Standard Error of Mean 1.112

3. Secondary Outcome: LS Mean of Change From Baseline in PGI-S From a Mixed Model for Repeated Measures
Description: Patient Global Impression - Severity (PGI-S) is participant reported assessment designed to evaluate the severity of their Parkinson's Disease. Scores range from 1 to 4 with 1 considered Normal and 4 considered Severe.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
score on a scale | 0.04 [-0.114 to 0.203] | 0.13 [-0.023 to 0.279] | 0.03 [-0.134 to 0.185] | -0.04 [-0.193 to 0.118]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of treatment; Test type: Superiority; p = 0.463, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.139 to 0.304], Standard Error of Mean 0.112
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.133, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.051 to 0.383], Standard Error of Mean 0.110
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.575, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.159 to 0.286], Standard Error of Mean 0.112

4. Secondary Outcome: LS Mean of Change From Baseline in CGI-S From a Mixed Model for Repeated Measures
Description: Clinician Global Impression - Severity (CGI-S) is clinician reported assessment designed to evaluate the severity of a participants Parkinson's disease. Scores range from 1 to 7 with 1 considered "Normal" and 7 considered "Among the most extremely ill patients".
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
score on a scale | -0.08 [-0.291 to 0.122] | 0.13 [-0.076 to 0.329] | -0.02 [-0.230 to 0.195] | 0.11 [-0.090 to 0.317]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 week of dosing; Test type: Superiority; p = 0.178, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.488 to 0.092], Standard Error of Mean 0.146
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.931, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.274 to 0.300], Standard Error of Mean 0.145
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.380, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.426 to 0.163], Standard Error of Mean 0.149

5. Secondary Outcome: LS Mean of Change From Baseline in MDS-UPDRS Part II From a Mixed Model for Repeated Measures
Description: Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Part II assesses activities of daily living as reported by the participant. Part II consists of 13 items with a total score ranging from 0 to 52. Each item is scored 0 (normal) to 4 (severe). Higher scores reflect increased severity of disease.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scale score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Scale score | 0.11 [-0.836 to 1.047] | -0.32 [-1.243 to 0.604] | -0.08 [-1.051 to 0.894] | 1.09 [0.157 to 2.020]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.144, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.98, 95% CI 2-sided [-2.308 to 0.342], Standard Error of Mean 0.669
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.036, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -1.41, 95% CI 2-sided [-2.720 to -0.096], Standard Error of Mean 0.662
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.089, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -1.17, 95% CI 2-sided [-2.514 to 0.180], Standard Error of Mean 0.680

6. Secondary Outcome: LS Mean of Change From Baseline in MDS-UPDRS Part III From a Mixed Model for Repeated Measures
Description: Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Part III is completed by clinician and assesses a participants motor function. Part III consists of 18 items with a total score ranging from 0 to 132. Each item is scored 0 (normal) to 4 (severe). Higher scores reflect increased severity of disease.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment Score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment Score | -0.04 [-2.381 to 2.309] | 2.14 [-0.161 to 4.438] | 2.20 [-0.216 to 4.620] | -0.21 [-2.534 to 2.112]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.916, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.18, 95% CI 2-sided [-3.127 to 3.477], Standard Error of Mean 1.668
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.158, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 2.35, 95% CI 2-sided [-0.921 to 5.621], Standard Error of Mean 1.652
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.157, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 2.41, 95% CI 2-sided [-0.941 to 5.768], Standard Error of Mean 1.694

7. Secondary Outcome: LS Mean of Change From Baseline in MDS-UPDRS Part I From a Mixed Model for Repeated Measures
Description: Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Part I assesses non-motor experiences of daily living. Part I is made up of two section with one rated by the investigator and another completed by the participant. Part I consists of 13 items with a total score ranging from 0 to 52. Each item is scored 0 (normal) to 4 (severe). Higher scores reflect increased severity of disease.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assesment Score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assesment Score | -0.93 [-1.842 to -0.028] | -1.03 [-1.919 to -0.133] | 0.22 [-0.716 to 1.161] | -0.26 [-1.159 to 0.638]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.297, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.67, 95% CI 2-sided [-1.952 to 0.602], Standard Error of Mean 0.645
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.233, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.77, 95% CI 2-sided [-2.032 to 0.500], Standard Error of Mean 0.639
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.464, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.48, 95% CI 2-sided [-0.818 to 1.783], Standard Error of Mean 0.657

8. Secondary Outcome: LS Mean of Change From Baseline in NMSS From a Mixed Model for Repeated Measures
Description: Non-Motor Symptom Score (NMSS) is a 30 question assessment completed by the clinician designed to evaluate the non-motor symptoms of Parkinson's disease. Scores range from 0 to 360 with higher scores reflect increasing severity of disease
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment score | 0.14 [-5.303 to 5.581] | 0.79 [-4.451 to 6.032] | 0.88 [-4.676 to 6.435] | -0.14 [-5.470 to 5.196]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.943, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.28, 95% CI 2-sided [-7.346 to 7.898], Standard Error of Mean 3.845
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.806, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.93, 95% CI 2-sided [-6.547 to 8.402], Standard Error of Mean 3.769
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.794, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 1.02, 95% CI 2-sided [-6.686 to 8.719], Standard Error of Mean 3.884

9. Secondary Outcome: LS Mean of Change From Baseline in CSBM Score From a Mixed Model for Repeated Measures
Description: The Complete Spontaneous Bowel Movement (CSBM) Diary is a participant-completed paper diary used to record bowel movement activity over a 7-day period. Each entry captures the date and time of the bowel movement, stool consistency (Bristol Stool Form Scale), and whether the bowel movement was spontaneous (no laxative or rescue medication within the previous 24 hours) and complete (a sensation of full evacuation).
  The weekly CSBM score is calculated as the total number of complete and spontaneous bowel movements recorded during the 7-day period. Rome IV criteria defines constipation as having less than 3 CSBMs per 7 day period. A decrease in CSBM score represents a decrease in bowel function.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of bowel movements per week
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Number of bowel movements per week | -0.04 [-0.963 to 0.875] | 0.30 [-0.588 to 1.189] | -0.11 [-1.012 to 0.794] | 0.85 [-0.062 to 1.767]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.173, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.90, 95% CI 2-sided [-2.193 to 0.400], Standard Error of Mean 0.654
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.393, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.55, 95% CI 2-sided [-1.828 to 0.725], Standard Error of Mean 0.644
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.141, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.96, 95% CI 2-sided [-2.246 to 0.323], Standard Error of Mean 0.648

10. Secondary Outcome: LS Mean of Change From Baseline in ESS From a Mixed Model for Repeated Measures
Description: The Epworth Sleepiness Scale is a self-administered questionnaire that measures a participant's general level of daytime sleepiness. Participants rate their likelihood of dozing off or falling asleep in eight common situations using a 4-point scale from 0 = would never doze to 3 = high chance of dozing. The total ESS score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment Score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment Score | -0.46 [-1.277 to 0.356] | -0.30 [-1.081 to 0.472] | -0.76 [-1.580 to 0.054] | -0.68 [-1.485 to 0.122]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.704, Mixed Models Analysis — Study not sized for efficacy; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.925 to 1.366], Standard Error of Mean 0.578
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.506, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.38, 95% CI 2-sided [-0.742 to 1.494], Standard Error of Mean 0.564
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.888, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.08, 95% CI 2-sided [-1.227 to 1.063], Standard Error of Mean 0.578

11. Secondary Outcome: LS Mean of Change From Baseline in SE-ADL From a Mixed Model for Repeated Measures
Description: Schwab and England Activies of Daily Living (SE-ADL) is a clinician administered assessment whereby participants assess their ability to complete routine daily activities on a scale from 0 to 100. The score is reported in increments of 10 with 100 representing normal ability to complete daily activities.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment Score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment Score | 0.02 [-0.001 to 0.038] | -0.00 [-0.019 to 0.018] | -0.00 [-0.023 to 0.017] | -0.02 [-0.040 to -0.002]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.004, Mixed Models Analysis — Study was not sized to evaluate efficacy; Mean Difference (Net) = 0.04, 95% CI 2-sided [0.013 to 0.067], Standard Error of Mean 0.014
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.125, Mixed Models Analysis — Study was not sized to evaluate efficacy; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.006 to 0.047], Standard Error of Mean 0.013
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.179, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.009 to 0.046], Standard Error of Mean 0.014

12. Secondary Outcome: LS Mean of Change From Baseline in PAGI-SYM From a Mixed Model for Repeated Measures
Description: The Patient Assessment of Upper Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) is a participant-reported questionnaire designed to assess the severity of upper gastrointestinal symptoms over the previous two weeks. The instrument includes 20 items. Each item is rated on a 6-point Likert scale from 0 = none to 5 = very severe, with higher scores indicating greater symptom severity. A total score is calculated as the mean of non-missing item responses.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment score | -0.04 [-0.179 to 0.089] | -0.02 [-0.154 to 0.109] | -0.09 [-0.229 to 0.050] | 0.05 [-0.083 to 0.183]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.321, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.283 to 0.094], Standard Error of Mean 0.095
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.444, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.259 to 0.114], Standard Error of Mean 0.094
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.154, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.332 to 0.053], Standard Error of Mean 0.097

13. Secondary Outcome: LS Mean of Change From Baseline in PAC-QoL From a Mixed Model for Repeated Measures
Description: The Patient Assessment of Constipation Quality of Life (PAC-QOL) is a participant-reported questionnaire that evaluates the impact of constipation and its treatment on quality of life over the previous two weeks. It consists of 28 items. Each item is rated on a 5-point Likert scale from 0 = not at all / very satisfied to 4 = extremely / very dissatisfied, depending on item phrasing. Scores are calculated as the mean of all non-missing items, with higher scores indicating greater negative impact on quality of life.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment Score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment Score | -0.03 [-0.173 to 0.120] | -0.17 [-0.310 to -0.027] | -0.13 [-0.277 to 0.023] | -0.03 [-0.177 to 0.111]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.950, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.199 to 0.212], Standard Error of Mean 0.104
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.189, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.338 to 0.067], Standard Error of Mean 0.102
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.374, Mixed Models Analysis; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.301 to 0.114], Standard Error of Mean 0.105

14. Secondary Outcome: LS Mean of Change From Baseline in PAGI-QoL From a Mixed Model for Repeated Measures
Description: The Patient Assessment of Upper Gastrointestinal Disorders Quality of Life (PAGI-QOL) is a validated, participant-reported questionnaire that assesses the impact of upper gastrointestinal symptoms on quality of life over the previous two weeks. The instrument includes 30 items. Each item is rated on a 6-point Likert scale from 0 = none of the time to 5 = all of the time. Scores are calculated as the mean of all non-missing items, with lower scores represent a greater negative impact on a participant's quality of life.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Assessment score
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 32 | 32 | 29 | 32
Assessment score | 0.07 [-0.014 to 0.150] | 0.06 [-0.023 to 0.139] | 0.06 [-0.030 to 0.141] | 0.05 [-0.029 to 0.135]
Statistical Analysis 1: Comparison: 50mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.803, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.101 to 0.131], Standard Error of Mean 0.058
Statistical Analysis 2: Comparison: 100mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.935, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.110 to 0.120], Standard Error of Mean 0.058
Statistical Analysis 3: Comparison: 200mg IkT-148009 (Risvodetinib); Change relative to placebo at 12 weeks of dosing; Test type: Superiority; p = 0.968, Mixed Models Analysis — Study not sized to evaluate efficacy; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.116 to 0.121], Standard Error of Mean 0.060

15. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 35 | 34 | 33 | 35
Participants | 19 | 21 | 21 | 21

16. Primary Outcome: Proportion of Those Randomized in Each Dosing Cohort Who Discontinued the Assigned Regimen Due to an Adverse Event
Time Frame: Baseline to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
Number analyzed (Participants) | 35 | 34 | 33 | 35
Participants | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Enrollment until the end of follow up (14 weeks post baseline visit)
Description: All adverse event recordings were done in compliance with ICH and FDA guidance
Arm/Group | 50mg IkT-148009 (Risvodetinib) | 100mg IkT-148009 (Risvodetinib) | 200mg IkT-148009 (Risvodetinib) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34 | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/34 | 1/33 | 1/35
Other Adverse Events (participants affected / at risk) | 19/35 | 21/34 | 21/33 | 21/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg IkT-148009 (Risvodetinib) (N=35) | 100mg IkT-148009 (Risvodetinib) (N=34) | 200mg IkT-148009 (Risvodetinib) (N=33) | Placebo (N=35)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related
Infection of Finger (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not Related
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg IkT-148009 (Risvodetinib) (N=35) | 100mg IkT-148009 (Risvodetinib) (N=34) | 200mg IkT-148009 (Risvodetinib) (N=33) | Placebo (N=35)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lipase Increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 5 (5)
Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye Swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular Discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Adverse drug reaction (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localized Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthopod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Post procedural erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood oestrogen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine leukocyte esterase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Action tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intention tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless leg syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Typical aura without headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disturbance in social behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnmbulism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Obstructive sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion of the Study and evaluation by Sponsor of all data from the Study, or upon early termination or abandonment of the Study, Institution and Investigator may publish or otherwise publicly disclose, for non-commercial purposes, Study Data .

DOCUMENTS (2):
  • Study Protocol (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT05424276/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT05424276/SAP_001.pdf